CLINICAL TRIAL: NCT03181867
Title: 18F-DCFPyL PET/CT in High Risk and Recurrent Prostate Cancer
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 170109; 17-C-0109
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01-16

CONDITIONS: Prostate Neoplasms; Prostatic Cancer; Prostate Cancer; Cancer Of Prostate; Metastatic Prostate Cancer
Keywords: Endorectal MRI; Imaging; PSMA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; Fluorodeoxyglucose F18; PSMA-11

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Localized High Risk (Experimental): 18F-DCFPyL PET/CT imaging, unlabeled PSMA-11 (optional) and possible prostatectomy
  Interventions: Drug: 18F-DCFPyL; Drug: PSMA-11
- 2/biochemical recurrence (bcr) (Experimental): 18F-DCFPyL PET/CT imaging, unlabeled PSMA-11 (optional)
  Interventions: Drug: 18F-DCFPyL; Drug: 18F-FDG; Drug: PSMA-11

INTERVENTIONS:
Drug: 18F-DCFPyL — Subjects will receive IV dose of 18F-DCFPyL by bolus injection. The maximum amount of injected active drug will be less than 4.02 mcg. The target administered activity will be 8 mCi.
Drug: 18F-FDG — Cohort 2 may receive a one-time 18F-FDG PET/CT after a positive 18F-DCPyL PET/CT. 18F FDG PET/CT imaging may be performed per clinical standard of care. FDG is administered at a dose of 10mCi intravenously. A whole-body PET/CT will be performed beginning post 18F FDG injection.
  Arms: 2/biochemical recurrence (bcr)
Drug: PSMA-11 — For up to 10 eligible patients from either cohort 1 or 2, an optional salivary gland blocking study may be performed in which a salivary gland is cannulated and injected with unlabeled DCFPyL or PSMA-11.

SUMMARY:
Background:

Prostate cancer is the second leading cause of cancer deaths in American men. When prostate cancer is confined to the prostate there is a high chance of cure. However, it is outside the prostate or comes back after treatment, additional therapy may be needed. Current methods of imaging prostate cancer are limited. Researchers want to see if a radiotracer called 18F-DCFPyL can identify prostate cancer in patients who have a high risk of cancer spreading outside the prostate or who have signs of recurrent cancer after treatment.

Objectives:

To see if the radiotracer 18F-DCFyL can help identify prostate cancer in the body before or after therapy.

Eligibility:

Men ages 18 and older who have prostate cancer that has been newly diagnosed, or has relapsed after radiation or surgery

Design:

Participants will be divided into 2 groups.

* Group 1 will be men with cancer that has been newly diagnosed as high risk by their doctor who are scheduled to have prostate removal surgery or undergo biopsy before radiation therapy.
* Group 2 will be men who have presumed prostate cancer relapse after prostate removal surgery or radiation therapy.

Both groups will have scans taken. Participants will lie still on a table in a machine that takes pictures of their body. 18F-DCFyL will be injected by intravenous (IV) line.

Participants will be contacted for follow-up after scans.

Participants in Group 1 may have surgery to remove their prostate gland or a biopsy to remove some prostate tissue. This procedure will be standard of care and is not a part of this study. They will also have an extra MRI scan of their prostate. For this, a tube, called an endorectal coil, will be placed in their rectum. Other tubes may be wrapped around the inside of their pelvis. A contrast agent will be given by IV.

Participants in Group 2 may also undergo an MRI of the pelvis and may have a biopsy of abnormalities found on the 18F-DCFyL scan.

Participants will have data about their prostate cancer collected for up to 1 year.

DETAILED DESCRIPTION:
Background:

* Prostate cancer (PCa) is the second leading cause of cancer death in American males.
* Patients with high risk but apparently localized disease are often understaged because disease beyond the prostate is not well detected and thus leads to overtreatment with prostatectomy
* Recurrence of PCa after surgery or radiation is very common and sometimes progresses to death.
* Early intervention for recurrence has been shown to be of benefit but current methods of localizing recurrence are either insensitive (CT), non-specific (MRI) or both (bone scan). Many prostate cancers express the prostate specific membrane antigen (PSMA) a transmembrane protein with NAALADase (N-acetylated-alpha-linked-acidic dipeptidase) and folate hydrolase enzymatic activity. PSMA is also expressed in angiogenesis but otherwise has limited expression in normal tissue.
* An initial test of 18F-DCFBC, a first-generation PET agent targeting PSMA, in patients with advanced local disease and biochemically recurrent prostate cancer demonstrated the potential of PET to detect sites of recurrence but it was hampered by excessive blood pool activity.
* (18)F-DCFPyL, a second generation PSMA PET agent, binds with high affinity to PSMA yet clears rapidly from the blood pool and thus, whole-body PET imaging with this agent, may provide a new tool in staging high risk cancers and detecting recurrent disease.

Primary Objective:

-To assess the ability of 18F-DCFPyL to accurately stage high-risk primary prostate cancer and detect sites of recurrent prostate cancer.

Eligibility:

* Age >=18 years old
* ECOG 0-2
* Histologically confirmed adenocarcinoma of the prostate
* Patients fit criteria for one of the following categories:

  * Cohort 1: known localized high risk prostate cancer (PSA >10, Gleason 8-10 or clinical stage >T2c) with evidence of disease on standard imaging

or

--Cohort 2: nonspecific or no evidence of disease on standard imaging modality AND biochemical prostate cancer relapse with a PSA > 0.2 ng/ml

Design:

* This is a single site study evaluating 18F-DCFPyL high-risk primary prostate cancer and recurrent prostate cancer.
* All subjects will undergo 18F-DCFPyL injection and whole body PET/CT imaging, performed 2 hours (+/- 15 minutes) post 18F-DCFPyL injection.
* Up to 10 eligible patients in either cohort 1 or 2 will receive an additional (18)F-DCFPyL PET/CT scan within 1 month of the first study immediately after unilateral salivary gland cannulation and an infusion of unlabeled DCFPyL or PSMA-11 into the cannulated gland.
* Patients from cohort 2 who have a positive 18F-DCFPyL PET/CT scan at any time may also have a one-time 18F-FDG PET/CT within 30 days of the positive 18F-DCFPyL PET/CT.
* All patients will undergo a standard of care, clinical multiparametric MRI in the NCI Molecular Imaging Clinic within 4 months of the PET scan.
* The patients will be followed yearly for 4 years by chart review, phone-call, email or any other NIH approved platform for PSA relapse and radiologic evidence of metastatic disease. Additional (18)F-DCFPyL might be performed during the subject s follow up period if there has been a considerable change in patient status (progression or response) based on PSA value, symptomatology, bone scan or CT findings.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years old.
* Eastern Cooperative Oncology Group (ECOG) Performance score of 0 to 2.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Histologically confirmed adenocarcinoma of the prostate.
* Patients (including those receiving androgen deprivation therapy) fit criteria for one of the following categories:

  * Cohort 1 known localized high risk prostate cancer (PSA >10, Gleason 8-10 or clinical stage >T2c) with evidence of disease on standard imaging, OR
  * Cohort 2 nonspecific or no evidence of disease on standard imaging modality AND biochemical prostate cancer relapse with a PSA greater than or equal to 0.2 ng/mL. Patients must be willing to undergo mandatory research biopsy
* Participants must be co-enrolled on a MIB, UOB, GMB or ROB protocol.
* The effects of 18F-DCFPyL on the developing human fetus are unknown. For this reason, individuals must agree to use adequate contraception with their partner (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 2 months after 18F-DCFPyL scan. Should a partner become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform the treating physician immediately.

EXCLUSION CRITERIA:

* Subjects for whom participating would significantly delay the scheduled standard of care therapy.
* Subjects with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results.
* Subjects with severe claustrophobia unresponsive to oral anxiolytics
* Other medical conditions deemed by the principal investigator (or associates) to make the subject unsafe/ineligible for protocol procedures.
* Subjects weighing greater than 350 lbs. (weight limit for scanner table), or unable to fit within the imaging gantry.
* Serum creatinine greater than 2 times the upper limit of normal.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2017-08-03 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the ability of 18F-DCFPyL to accurately stage high-risk primary prostate cancer and detect sites of recurrent prostate cancer | 12 months
  Correlation between 18F-DCFPyL scanning and accurately staging of high-risk primary prostate cancer and detection of sites of recurrent prostate cancer.

SECONDARY OUTCOMES:
Evaluate the distribution of 18F-DCFPyL uptake in prostate cancer patients with biochemical relapse (site of recurrence unknown) as a function of PSA value | 12 month
  PSA value of the distribution of 18F-DCFPyL uptake in prostate cancer patients with biochemical relapse
Compare the distribution of 18F-DCFPyL uptake with multiparametric MRI and whole mount histopathology in patients undergoing prostatectomy | 12 month
  Correlation between the distribution of 18F-DCFPyL uptake and multiparametric MRI and whole mount histopathology in patients undergoing prostatectomy
Compare focal 18F-DCFPyL uptake with focal abnormalities identified on standard of care imaging | 12 month
  Correlation between focal 18F-DCFPyL uptake and focal abnormalities identified on standard of care imaging

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Choyke, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Chen Y, Pullambhatla M, Foss CA, Byun Y, Nimmagadda S, Senthamizhchelvan S, Sgouros G, Mease RC, Pomper MG. 2-(3-1-Carboxy-5-[(6-[18F]fluoro-pyridine-3-carbonyl)-amino]-pentyl-ureido)-pentanedioic acid, [18F]DCFPyL, a PSMA-based PET imaging agent for prostate cancer. Clin Cancer Res. 2011 Dec 15;17(24):7645-53. doi: 10.1158/1078-0432.CCR-11-1357. Epub 2011 Oct 31. PMID 22042970
- [Background] Cho SY, Gage KL, Mease RC, Senthamizhchelvan S, Holt DP, Jeffrey-Kwanisai A, Endres CJ, Dannals RF, Sgouros G, Lodge M, Eisenberger MA, Rodriguez R, Carducci MA, Rojas C, Slusher BS, Kozikowski AP, Pomper MG. Biodistribution, tumor detection, and radiation dosimetry of 18F-DCFBC, a low-molecular-weight inhibitor of prostate-specific membrane antigen, in patients with metastatic prostate cancer. J Nucl Med. 2012 Dec;53(12):1883-91. doi: 10.2967/jnumed.112.104661. PMID 23203246
- [Background] Szabo Z, Mena E, Rowe SP, Plyku D, Nidal R, Eisenberger MA, Antonarakis ES, Fan H, Dannals RF, Chen Y, Mease RC, Vranesic M, Bhatnagar A, Sgouros G, Cho SY, Pomper MG. Initial Evaluation of [(18)F]DCFPyL for Prostate-Specific Membrane Antigen (PSMA)-Targeted PET Imaging of Prostate Cancer. Mol Imaging Biol. 2015 Aug;17(4):565-74. doi: 10.1007/s11307-015-0850-8. PMID 25896814
- [Derived] Rowe LS, Harmon S, Horn A, Shankavaram U, Roy S, Ning H, Lindenberg L, Mena E, Citrin DE, Choyke P, Turkbey B. Pattern of failure in prostate cancer previously treated with radical prostatectomy and post-operative radiotherapy: a secondary analysis of two prospective studies using novel molecular imaging techniques. Radiat Oncol. 2021 Feb 10;16(1):32. doi: 10.1186/s13014-020-01733-x. PMID 33568190
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-C-0109.html